CLINICAL TRIAL: NCT00100568
Title: A Pilot Study of Safety, Effectiveness, and Adherence of Lamivudine/Zidovudine and Efavirenz (3TC/ZDV + EFV) to Treat HIV-1 Infection in Senegal
Brief Title: Efavirenz and Lamivudine/Zidovudine for Treatment-Naive HIV Infected Adults in Senegal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Initiative Senegalaise d'Acces aux Antiretroviraux (ISAARV) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIPRA-SN-001; SN-CIPRA-001; 10412 (Registry Identifier: DAIDS-ES); NCT00738465 (obsolete NCT alias)
Record Dates: First submitted 2005-01-03; First posted 2005-01-04 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-09

CONDITIONS: HIV Infections
Keywords: Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — efavirenz; lamivudine, zidovudine drug combination

ARMS (1):
- 1 (Experimental): All participants will be given an ARV regimen of lamivudine/zidovudine and efavirenz at study entry. If toxicity or treatment failure occurs, some participants may require changes in their ARV regimens.
  Interventions: Drug: Efavirenz; Drug: Lamivudine/zidovudine

INTERVENTIONS:
Drug: Efavirenz — 600 mg tablet taken orally daily
  Other Names: EFV
Drug: Lamivudine/zidovudine — 150mg lamivudine/300mg zidovudine tablet taken orally twice daily
  Other Names: 3TC/ZDV

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of the anti-HIV drugs efavirenz and lamivudine/zidovudine given to treatment-naive HIV-infected people in Dakar, Senegal.

DETAILED DESCRIPTION:
Despite a relatively low prevalence of HIV infection, all HIV subtypes have been documented in Senegal. Data on mutations that confer resistance to antiretroviral (ARV) drugs are limited to HIV subtype B; adherence data are also limited. The study will evaluate the safety and efficacy of an ARV regimen given to treatment-naive HIV infected adults and adolescents. The study will also examine the characteristics of virologic failure and adherence in this treatment group. Participants will be recruited at two sites in Dakar, Senegal.

This study will last 96 weeks. At study entry, all participants will be given an ARV regimen of lamivudine/zidovudine twice daily and efavirenz once daily. If toxicity or treatment failure occurs, some participants may require changes in their ARV regimens. There will be 14 study visits during the study; a physical exam, blood collection, and sociodemographic and medication history assessments will occur at each visit. Participants will also be asked to complete quality-of-life and adherence questionnaires. An off-study visit will occur at approximately one month after Week 96, with assessments and procedures similar to visits during the study.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected
* Have never taken ARV drugs
* CD4 count of 200 cells/mm3 or less within 30 days of study entry if asymptomatic OR CD4 count of 350 cells/mm3 or less within 60 days of study entry if CDC Category A or B clinical condition present OR clinical diagnosis of AIDS, regardless of CD4 count
* Willing to stay in the study area for the duration of the study
* Willing to use acceptable forms of contraception

Exclusion Criteria:

* HIV-2 infected
* Systemic chemotherapy (except interferon) within 6 months prior to study entry
* Current drug or alcohol abuse that, in the opinion of the investigator, may interfere with the study
* Serious illness, including any active AIDS-defining infection, active tuberculosis, malaria, or any illness requiring systemic treatment or hospitalization. People who have completed therapy or are clinically stable on therapy for at least 14 days prior to study entry are not excluded.
* Serious psychiatric problems within 60 days of study entry, including depression, suicidal thoughts or attempts, aggressive behavior, or psychosis-like symptoms
* Have taken certain medications within 30 days of study entry
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2006-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Virologic efficacy, defined as HIV-1 viral load less than 200 copies/ml | Through Week 24
Treatment-related toxicity of Grade 3 or higher as measured by development of drug-related toxicities severe enough to warrant dose modification, interruption, or permanent discontinuation | Through Week 24

SECONDARY OUTCOMES:
Virologic efficacy | At Weeks 48 and 96
Treatment related toxicity | At Weeks 48 and 96
Virologic failure, defined as HIV-1 viral load greater than 1,000 copies/ml | Throughout study
CD4 counts and HIV-1 RNA viral load | Throughout study
First new or recurrent AIDS-defining event (as defined by the CDC Expanded AIDS Surveillance Case definition) or death | Throughout study
Treatment discontinuation, defined as premature discontinuation of participation in the study, failure to take ARV therapy for 8 or more consecutive weeks, or to switch to another ARV regimen for any reason during the full course of the study | Throughout study
Genotypic resistance measured by at least 1 genotypic mutation associated with resistance among subjects with a confirmed virologic failure (as described previously) and evaluation of genotypic drug resistance patterns | At Weeks 24 and 96
Treatment adherence, defined by 95% or greater of prescribed pills taken | Throughout study
Quality of life as measured by items and patterns of responses to the FAHI questionnaire | Throughout study
HIV-1 DNA and RNA measurements | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Souleymane Mboup, PharmD, Study Chair — Laboratoire de Bacteriologic et de Virologie, Hospital Le Dantec Avenue Pasteur
Locations (2):
- Senegal (2):
  - Centre National Hospitalier de Fann, Dakar CIPRA CRS, Dakar
  - Institut d'Hygiène Sociale, Dakar CIPRA CRS, Dakar

REFERENCES:
- [Background] Meda N, Ndoye I, M'Boup S, Wade A, Ndiaye S, Niang C, Sarr F, Diop I, Carael M. Low and stable HIV infection rates in Senegal: natural course of the epidemic or evidence for success of prevention? AIDS. 1999 Jul 30;13(11):1397-405. doi: 10.1097/00002030-199907300-00018. PMID 10449294
- [Background] DeJesus E, Herrera G, Teofilo E, Gerstoft J, Buendia CB, Brand JD, Brothers CH, Hernandez J, Castillo SA, Bonny T, Lanier ER, Scott TR; CNA30024 Study Team. Abacavir versus zidovudine combined with lamivudine and efavirenz, for the treatment of antiretroviral-naive HIV-infected adults. Clin Infect Dis. 2004 Oct 1;39(7):1038-46. doi: 10.1086/424009. Epub 2004 Sep 10. PMID 15472858